CLINICAL TRIAL: NCT06213376
Title: Intensive MIT Paired With Video Feedback for Motor Speech Disorders and Aphasia
Brief Title: MIT Intensive Treatment Study
Acronym: MITTXS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nevada State University (Other)
Responsible Party: Principal Investigator, Andre Lindsey, Assistant Professor of Speech Pathology, Nevada State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2312-0370
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Aphasia; Motor Speech
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Intervention Model Description: Single-subject experimental design
Masking Description: Independent Raters will be used to examine non-standardized outcomes at benchmark time points.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): 20 sessions/4 weeks:
  Video Feedback:
  S1) Participant (P1) views recording of previous session with the clinician & judges whether the production is intelligible.
  S2) S1 & the clinician identifies changes in motor movements that are influencing performance.
  S3+S4) S1+S2 & given support from the clinician, P1 identifies techniques improving intelligibility & modifies behavior accordingly.
  MIT (Albert et al., 1973; Helm-Estabrooks et al., 2014):
  Humming - Clinician introduces the target phrase by showing a visual cue, humming the phrase, then intoning the phrase while P1 taps left-hand.
  Simultaneous production with melody - The Clinician and P1 melodically produce the target phrase & tap together.
  Simultaneous melodic production accompanied by gradual reduction of clinician support.
  Immediate repetition response to probe question - Following P1's successful repetition, the clinician melodically produces a question and P1 melodically produces the target.
  Interventions: Behavioral: Melodic Intonation Therapy; Behavioral: Video Feedback Performance Review

INTERVENTIONS:
Behavioral: Melodic Intonation Therapy — Melodic Intonation Therapy uses intonation and melody to aid individuals with aphasia with producing words.
Behavioral: Video Feedback Performance Review — Participant will view recording to judge correct and incorrect productions of trained words and to identify motor techniques increasing intelligibility

SUMMARY:
This study is examining the use of intensive melodic intonation therapy and video feedback as a means of aiding individuals with nonfluent aphasia and co-occurring motor speech impairments. Individuals with nonfluent aphasia have difficulty with language, particularly with word retrieval.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English speakers
* Sustained a left-hemisphere stroke
* Presents with language and motor speech impairments

Exclusion Criteria:

* • History of learning disability prior to accident (per patient report)

  * Uncorrected auditory or visual impairments
  * Not meeting the criteria of stroke
  * Failure to provide evidence of stroke diagnosis (medical record history)
  * History of psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Intelligibility | From enrollment to 4 weeks post treatment
  Intelligibility as measured by percentage of consonants correct and by targets produced on trained and untrained stimuli. 20 trained and 20 untrained speech phrases that are relevant to the client (measured during reading and repetition tasks)

SECONDARY OUTCOMES:
Apraxia Battery for Adults | Baseline and one week following the end of treatment
  A test to measure the presence and severity of apraxia in adults
Assessment of Intelligibility of Dysarthria Speech | Baseline and one week following the end of treatment
  A tool for quantifying single-word intelligibility, sentence intelligibility, and speaking rate of adult speakers with dysarthria
Longer Connected Speech Assessment | Baseline and one and four weeks following the end of treatment
  Change in Performance on Rainbow Passage- A public domain paragraph frequently used by speech-language pathologists to gather a speech sample of all phonemes for American English
Quality of Life with Dysarthria (QOLdys) | Baseline and four weeks following treatments.
  A reliable and valid tool to assess quality of life for patients with dysarthria.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Lindsey, PhD, Principal Investigator — Nevada State University
Locations (1):
- Nevada State University, Henderson, Nevada, United States

REFERENCES:
- [Background] Albert ML, Sparks RW, Helm NA. Melodic intonation therapy for aphasia. Arch Neurol. 1973 Aug;29(2):130-1. doi: 10.1001/archneur.1973.00490260074018. No abstract available. PMID 4717723
- [Background] Helm-Estabrooks, N., Albert, M. L., & Nicholas, M. (2014). Manual of aphasia and aphasia therapy (3rd ed.). Austin, TX: Pro-Ed
- [Background] Zumbansen A, Peretz I, Hebert S. Melodic intonation therapy: back to basics for future research. Front Neurol. 2014 Jan 28;5:7. doi: 10.3389/fneur.2014.00007. eCollection 2014. PMID 24478754